CLINICAL TRIAL: NCT01103427
Title: Mobile Text Messaging as an Adjunct Function to an Internet-based Smoking Cessation Intervention Implemented in the General Population and in a Health Care Setting
Brief Title: Usefulness of Supportive SMS in Addition to an Internet Based Quit Smoking Program (Www.Slutta.no)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tromso (Other)
Collaborators: The Royal Norwegian Ministry of Health (Other); University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TFP-743-08
Record Dates: First submitted 2010-04-13; First posted 2010-04-14 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Smoking Cessation; Smoking
Keywords: smoking cessation; telemedicine; smoking; prevention intervention; internet-based; text messages; behavioral
MeSH Terms: conditions — Smoking Cessation; Smoking; Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Internet-based coaching . (Active Comparator): Arm 1. Those in the "active comparator arm" will benefit from automated internet-based coaching. The subjects will be recruited from the general population reporting not to be associated with the University Hospital of North Norway and randomized to arm 1 or 2.
  Interventions: Device: Internet-based behavioral coaching
- SMS based coaching (Experimental): Arm 2. The subjects will receive automated "coaching"by SMS.The subjects will be recruited from the general population reporting not to be associated with the University Hospital of North Norway and randomized to arm 1 or 2.
  Interventions: Device: SMS based coaching
- SMS coaching UNN recruited (Experimental): Arm 3.The subjects will be recruited from those reporting to be associated with the University Hospital of North Norway and randomized to arm 3 or 4.
  Interventions: Device: SMS coaching - UNN recruited
- Craving/Panic function. UNN recruited (Experimental): Arm 4. The subjects will in addition to the automated "coaching"by SMS get a SMS panic/craving function. The subjects will be recruited from subjects reporting to be associated with the University Hospital of North Norway and randomized to arm 3 or 4.
  Interventions: Device: SMS craving function - UNN recruited

INTERVENTIONS:
Device: Internet-based behavioral coaching — Those in the "active comparator arm" will benefit from automated coaching by e-mails with advice, information and support for smoking cessation. These e-mails will be adapted to their personal profile.
  Other Names: slutta.no
  Arms: Internet-based coaching .
Device: SMS based coaching — Those in the experimental SMS based coaching arm will benefit from automated coaching by SMS with advice, information and support for smoking cessation. These SMS's will be adapted to their personal profile.
  Other Names: slutta.no
  Arms: SMS based coaching
Device: SMS coaching - UNN recruited — Those in the experimental SMS based coaching arm- UNN recruited - will benefit from automated coaching by SMS with advice, information and support for smoking cessation. These SMS's will be adapted to their personal profile.
  Other Names: slutta.no/unn
  Arms: SMS coaching UNN recruited
Device: SMS craving function - UNN recruited — Those in the experimental SMS based craving/panic function arm - will in addition to the automated coaching by SMS have a panic/craving SMS function. Thus by sending a SMS they will receive instant advise and support for smoking cessation by SMS.
  Other Names: slutta.no/unn
  Arms: Craving/Panic function. UNN recruited

SUMMARY:
The purpose of the study is to investigate the effectiveness of a smoking cessation intervention delivered through a technological web based platform (www.slutta.no) with or without a supportive SMS function.

DETAILED DESCRIPTION:
The study has two arms and are conducted in Norwegian. Users who registered with a new username on www.slutta.no, after study start May 12th 2010 and before November 1st 2012, are eligible. All phases of the trial, from randomization and informed consent procedures to data collection, are automated and conducted online. The following inclusion criteria are used: age 16 years or older, access to a mobile phone with a Norwegian phone number and they must submit an informed consent form.

ELIGIBILITY:
Inclusion Criteria (all arms):

* Aged 16 and older
* Current smoker: Willing to quit smoking within the next 12 weeks
* Former smokers; Having quit smoking within the previous six months
* Having a regular access to Internet
* Having a personal e-mail address
* Having a personal mobile cell phone with a Norwegian number
* Given informed consent
* Can read and understand Norwegian
* Reporting no association with the University Hospital of North Norway (arm1&2)
* Reporting an association with the University Hospital of North Norway (arm3&4)

Exclusion Criteria:

* Less than 16 years of age
* No personal e-mail address
* No personal mobile cell phone
* Not able to give the informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4300 (Actual)
Dates: Start 2010-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Comparison of the percentage of abstinent people between the arms of the trial,1,3,6 and 12 months after self-reported smoking cessation date | 30 months after inclusion
  The investigators will compare the percentage of smokers who successfully quit. Point prevalence abstinence will be measured (not smoking, event a puff, in the week preceding the questioning).

SECONDARY OUTCOMES:
Comparison between the arms of the trial regarding visits, time logged in, used elements of the website and overall adherence period. | 30 months after inclusion
  Number of visits to the website, time logged in, used elements of the website and adherence to the program will be measured utilizing the registrations on the server.
Comparison between the arms of the trial regarding satisfaction with website and mobile text messages at the time of the 4 questionnaires | 30 months after inclusion
  The 4 questionnaires comprise questions regarding satisfaction with website or text messages for the different arms depending om which device they have been utilizing.
28 days of continuous smoking prevalence at 6 months after selfreported smoking cessation date | 6 months after selfreported smoking cessation date
  Comparison between the four arms regarding self-reported 28 days continuous smoking abstinence through questionnaire
Selfreported involvement in any vehicle crashes during the last 6 months | 6 months after selfreported smoking cessation date
  Involvement in any vehicle crashes (this is the only rare adverse health effects of using a mobile phone)during the 6 months after selfreported smoking cessation date.

CONTACTS AND LOCATIONS:
Overall Officials: Inger T Gram, MD, PhD, Principal Investigator — University of Tromso; Bjørn Engum, Study Director — University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Norway

REFERENCES:
- [Derived] Gram IT, Larbi D, Wangberg SC. Comparing the Efficacy of an Identical, Tailored Smoking Cessation Intervention Delivered by Mobile Text Messaging Versus Email: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Sep 27;7(9):e12137. doi: 10.2196/12137. PMID 31573935